CLINICAL TRIAL: NCT06429072
Title: Integration of Mindfulness and Acupuncture After Spine Surgery: Aim 2
Brief Title: Integration of Mindfulness and Acupuncture After Spine Surgery
Acronym: I-MASS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pro00114814
Record Dates: First submitted 2024-03-04; First posted 2024-05-24 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-07

CONDITIONS: Single Level Spinal Fusion; Discetomy; Laminectomy
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- I-MASS Program plus Enhanced Education (Experimental)
  Interventions: Behavioral: Mindfulness training; Other: Acupuncture; Behavioral: Enhanced education
- Enhanced Education Intervention Only (Active Comparator)
  Interventions: Behavioral: Enhanced education

INTERVENTIONS:
Behavioral: Mindfulness training — • I-MASS begins with one introductory telephone call by a mindfulness coach within 1 week of the patient scheduling surgery to introduce the participant to the Pattern Health app, discuss the benefits of combining mindfulness and acupuncture, discuss how to access the Healthwise educational content, and lead a brief (~10 min) mindfulness exercise, as desired. Thereafter, participants will complete 4 self-directed mindfulness modules through the Pattern Health app (1 prior to surgery, 3 following surgery). Each mindfulness module is anticipated to last one week and includes a short (4-5 min) introductory video, daily sessions comprised of a 6-8 min guided mediation, and interactive suggestions for how to apply mindfulness within a daily routine (~10-12 min total per daily session).
  Arms: I-MASS Program plus Enhanced Education
Other: Acupuncture — This arm also includes up to 8 total acupuncture treatments (1 prior to surgery and up to 7 treatments in the 12 weeks after surgery). Auricular acupuncture will be the preferred form of acupuncture used. This technique involves inserting tiny needles in specific areas of the outer ear to target points believed to influence pain. If participants are unable to tolerate auricular acupuncture, they will have the option to receive peripheral acupuncture.
  Arms: I-MASS Program plus Enhanced Education
Behavioral: Enhanced education — • The program consists of education prior to and after surgery for all participants. All of the educational material is delivered via the Pattern Health App. All educational content is from the Healthwise.net Duke Health Library (https://www.healthwise.net/dukehealth/Content) and is carefully selected with input by surgeons to be delivered during the appropriate phase of recovery. Education is in the form of short reading materials or videos, all designed to help safely and effectively recover from surgery. Educational topics include learning how to lift and sit when experiencing pain, proper precautions following surgery, how to ease back into daily activities following surgery, and ways to self-manage pain.

SUMMARY:
The Integration of Mindfulness and Acupuncture for individuals undergoing Spine Surgery (I-MASS) is a novel combination of integrative treatments to improve post-surgical recovery.

This is a single-site, two-arm randomized feasibility and acceptability pilot trial of the I-MASS program plus enhanced patient education compared to enhanced patient education alone in patients undergoing spine surgery. Outcomes data will come from a combination of passive electronic health record data augmented with patient-reported data collected through the Pattern Health app (the mHealth platform used for delivering mindfulness training and collecting data). Outcomes will focus on feasibility and acceptability of I-MASS, feasibility of recruitment and retention strategies, and data collection procedures through both the Pattern Health app and electronic health record. Feasibility will be supported by mindfulness module completion rates, acupuncture visits attended, participant retention, and questionnaire completion rates. Acceptability will be supported by patient-reported satisfaction, acceptability and usability thresholds.

DETAILED DESCRIPTION:
Participants will be randomized to one of two study arms: 1) the I-MASS program plus enhanced education or 2) the enhanced education intervention only.

I-MASS program plus enhanced education (Intervention) Arm: This arm begins with one introductory telephone call by a mindfulness coach within 1 week of the patient scheduling surgery to introduce the participant to the Pattern Health app, discuss the benefits of combining mindfulness and acupuncture, discuss how to access the Healthwise educational content, and lead a brief (~10 min) mindfulness exercise, as desired. Thereafter, participants will complete 4 self-directed mindfulness modules through the Pattern Health app (1 prior to surgery, 3 following surgery). The modules will include a guided series of videos, audio files and interactive text features. Each week-long module includes daily sessions comprised of a short (4-5 min) background video, a 6-8 min guided mediation (users could choose either a female or male voice) and interactive suggestions for how to apply mindfulness within their daily routine (~10-12 min total per session). The pre-operative training (module 1) focuses on developing an awareness of breath, which is a fundamental mindfulness technique. Following surgery, participants will initiate training module 2, building awareness of body systems, followed by modules 3 and 4 over the subsequent 2 weeks. Automated activity reminders in the app will alert the participant to complete the daily session. Each module builds upon skills learned in the previous module and participants are encouraged to continue using learned skills and resources within the app after completion of the modules.

The initial acupuncture session will occur within one week prior to surgery. The second acupuncture session will occur within the first week following surgery. Afterwards, participants will receive acupuncture in participating community outpatient clinics for up to 8 sessions total within 12 weeks of surgery. The investigators will allow flexibility in scheduling these visits with a window of 5-10 days between acupuncture sessions. Acupuncturists will also be trained to facilitate discussion about mindful awareness and non-judgmental thoughts regarding pain, giving participants an opportunity to reflect on their experiences during the acupuncture session. Auricular acupuncture will be the preferred form of acupuncture used. If participants are unable to tolerate auricular acupuncture, they will have the option to receive peripheral acupuncture.

The program consists of enhanced education prior to and after surgery for all participants. All of the educational material is delivered via the Pattern Health App. All educational content is from the Healtwise.net Duke Health Library (https://www.healthwise.net/dukehealth/Content) and is carefully selected with input by surgeons to be delivered during the appropriate phase of recovery. Educational topics include learning how to lift and sit when experiencing pain, proper precautions following surgery, how to ease back into daily activities following surgery, and ways to self-manage pain. Education is in the form of short reading materials or videos, all designed to help safely and effectively recover from surgery.

Enhanced Education Arm: Participants in this arm will receive an introductory call from study staff to introduce the participant to the Pattern Health app, discuss how to access the Healthwise educational content, and answer any questions about the program. They will then receive the same course of enhanced educational material as the Intervention arm in the Pattern Health app.

All trial participants will not be prevented from receiving any other care deemed necessary by their health care team and surgeon. This program is designed to complement their usual care, not replace it. Participant involvement with the study will be complete at 3 months following surgery. All follow-up questionnaires will be administered through the Pattern Health app for participants in both study arms.

ELIGIBILITY:
Inclusion Criteria:

1. undergoing single level fusion, discectomy or laminectomy of the cervical or lumbar spine for management of pain
2. 18 years of age or older
3. has access to a smartphone or mobile device (with android or iOS operating system) and internet to complete training and questionnaires.

Exclusion Criteria:

1. have conditions making consent, follow-up data collection and/or use of the intervention prohibitive (e.g., Non-English speaking, serious psychiatric conditions [i.e., schizophrenia], traumatic brain injury, or dementia-type illness)
2. undergoing surgery for neoplastic disease
3. current daily opioid use greater than 100mg morphine equivalents
4. unable to receive acupuncture due to injury, infection, or other contraindication to the use of needles at acupuncture sites
5. not possible to attend outpatient clinic for AA follow-up (e.g., from out-of-state)
6. currently practicing mindfulness or receiving acupuncture
7. in Hospice, receiving palliative care.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-08-15 (Actual); Primary Completion 2025-10-15 (Actual); Study Completion 2025-10-15 (Actual)

PRIMARY OUTCOMES:
Client Satisfaction Questionnaire (CSQ-8) | up to 3 months post-surgery
  The CSQ-8 assesses credibility and satisfaction with health-related services (8 items, 4-point Likert, with higher scores indicating higher credibility/satisfaction).
Recruitment | up to 3 months post-surgery
  Percentage of contacted patients that are eligible and agree to participate
Data Collection | up to 3 months post-surgery
  Percentage of participants who complete self-report follow-up questionnaires at each of the 4 timepoints.
Number of completed acupuncture visits | up to 3 months post-surgery
  Percentage of acupuncture visits completed out of 8 possible visits
Number of completed mindfulness modules | up to 3 months post-surgery
  Percentage of completed mindfulness modules out of 4 possible in the Pattern Health app

SECONDARY OUTCOMES:
PROMIS-29 v2. 0 | Baseline (prior to surgery), 2weeks, 6weeks, 3 months post-surgery
  This profile assesses pain intensity using a single 0-10 numeric rating item and seven health domains (physical function, fatigue, pain interference, depressive symptoms, anxiety, ability to participate in social roles and activities, and sleep disturbance) using four items per domain and a one-item measure of pain intensity. This measure will be used to assess feasibility of data collection, no formal comparisons will be made across treatment arms.
Daily Pain Intensity | week before surgery, for 2 weeks after surgery
  Daily pain intensity during the week prior to surgery and for two weeks following surgery will be measured with the following two questions: 1) Please rate your worst pain in the last 24 hours on a scale from 0 (no pain) to 10 (worst possible pain), and 2) Please rate your average pain in the last 24 hours on a scale from 0 (no pain) to 10 (worst possible pain). These measures will be used to assess feasibility of data collection, no formal comparisons will be made across treatment arms.
SPARE Fear Avoidance Short-form | Baseline (prior to surgery) , 2weeks, 6weeks, 3 months post-surgery
  The SPARE-FA short form is a 4 item questionnaires that measures characteristics of pain-related fear avoidance, catastrophizing, and kinesiophobia. This measure will be used to assess feasibility of data collection, no formal comparisons will be made across treatment arms.
Medication Prescriptions | Baseline (prior to surgery) , 2weeks, 6weeks, 3 months post-surgery
  We will collect self-reported information on medication prescriptions for pain (e.g., Opioids, Benzodiazepines, Gabapentin/Neurontin, NSAIDs) at baseline, 6 weeks, and 3 months. We will also collect self-reported pain medication use daily during the first 2 weeks following surgery. This measure will be used to assess feasibility of data collection, no formal comparisons will be made across treatment arms.
Number of hospital readmission's related to spine surgery | up to 3 months post-surgery
  ADT alerts in the Epic EHR and periodic chart reviews through 3 months. This measure will be used to assess feasibility of data collection, no formal comparisons will be made across treatment arms.
Number of emergency room visits related to Spine. | up to 3 months post-surgery
  ADT alerts in the Epic EHR and periodic chart reviews through 3 months. This measure will be used to assess feasibility of data collection, no formal comparisons will be made across treatment arms.

CONTACTS AND LOCATIONS:
Overall Officials: Trevor Lentz, PhD, Principal Investigator — Duke University
Locations (1):
- Duke Sports Science Institute, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2025-03-17): https://cdn.clinicaltrials.gov/large-docs/72/NCT06429072/ICF_000.pdf